CLINICAL TRIAL: NCT01128933
Title: Prognostic Value of Renal Fractional Flow Reserve in Hypertensive Patients With Renal Artery Stenosis Qualified to Renal Artery Stenting
Brief Title: Renal Fractional Flow Reserve in Renal Artery Stenting
Acronym: PREFFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Jacek Kadziela, Institute of Cardiology, Warsaw, Poland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2P05B02530
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Renal Artery Stenosis; Hypertension
Keywords: Fractional flow reserve; Revascularization; Prognosis; Hemodynamics; Hypertension
MeSH Terms: conditions — Renal Artery Obstruction; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypertensive patients (Experimental): Hypertensive patients with at least moderate renal artery stenosis
  Interventions: Procedure: Renal artery stenting

INTERVENTIONS:
Procedure: Renal artery stenting

SUMMARY:
The purpose of the study is to determine potential utility of renal fractional flow reserve in prognosis predicting after renal stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* At least moderate (60% or more) renal artery stenosis with atheromatic appearance in angiography
* Hypertension defined according to WHO criteria
* Age 18-75 years
* Signed informed consent obtained

Exclusion Criteria:

* Bilateral renal artery stenosis or significant renal artery stenosis in solitary kidney
* Contraindications to percutaneous renal angioplasty with stenting
* Atrophy of the kidney supplied with stenosed artery
* Other well known secondary reason for hypertension
* Chronic heart failure NYHA II-IV
* Significant valvular heart disease qualified for surgery
* Persistent atrial fibrillation
* Renal failure with GFR below 30ml/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure improvement | 6 months

SECONDARY OUTCOMES:
Kidney function preservation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kadziela, MD,PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Adam Witkowski, Prof, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Andrzej Januszewicz, Prof, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Derived] Kadziela J, Prejbisz A, Michalowska I, Adamczak M, Warchol-Celinska E, Pregowska-Chwala B, Januszewicz M, Wiecek A, Januszewicz A, Witkowski A. Relationship between hemodynamic parameters of renal artery stenosis and the changes of kidney function after renal artery stenting in patients with hypertension and preserved renal function. Blood Press. 2015 Feb;24(1):30-4. doi: 10.3109/08037051.2014.958304. Epub 2014 Sep 30. PMID 25268986
- [Derived] Kadziela J, Januszewicz A, Prejbisz A, Michalowska I, Januszewicz M, Florczak E, Kalinczuk L, Norwa-Otto B, Warchol E, Witkowski A. Prognostic value of renal fractional flow reserve in blood pressure response after renal artery stenting (PREFER study). Cardiol J. 2013;20(4):418-22. doi: 10.5603/CJ.2013.0101. PMID 23913461
- See also: Web page of Institute of Cardiology, Warsaw — http://www.ikard.pl